CLINICAL TRIAL: NCT02998632
Title: The Effect of Posterior Mandibular Ridge Augmentation Using Mineralized Plasmatic Matrix Versus Autogenous Bone Graft on Implant Body Stability: A Randomized Clinical Trial Comparative Study
Brief Title: Posterior Mandibular Ridge Augmentation Using Mineralized Plasmatic Matrix Versus Autogenous Bone Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel-Sattar, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC - CU - 2016 - 11 - 165
Record Dates: First submitted 2016-12-02; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Bone Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional (Experimental): Patients will receive 2 gm of amoxicillin 1 hour before surgery. Mouthwash 0.12% chlorhexidine solution for 30 seconds immediately before surgery.
  Inferior alveolar nerve block and long buccal nerve anesthesia using articane HCl 4% with 1:100,000 adrenaline local anesthetic solution.
  Flap will be reflected in intraoral donor site to completely expose bone. Autogenous bone graft will be obtained and will be ground. MPM (Mineralized plasmatic matrix) will be prepared. Implant fixture/s will be inserted. Uncovered fixture threads and bone defect will be covered by MPM. Osstell will be used to measure fixture primary stability in ISQ units. Sutures will be placed. Sutures will be removed 7 days later. Immediate postoperative CBCT will be performed. Antibiotic (combination of 500mg amoxicillin and 125mg clavulanic acid) and analgesic and anti-inflammatory (Ibuprofen 600mg) will be prescribed.
  Interventions: Procedure: Mineralized plasmatic matrix for bone augmentation
- Comparator (Active Comparator): Patients will receive 2 gm of amoxicillin 1 hour before surgery. Mouthwash 0.12% chlorhexidine solution for 30 seconds immediately before surgery.
  The patient will receive inferior alveolar nerve block and long buccal nerve anesthesia using articane HCl 4% with 1:100,000 adrenaline local anesthetic solution Flap will be reflected in intraoral donor site to completely expose bone. Autogenous bone graft will be obtained and will be ground. Implant fixture/s will be inserted. Uncovered fixture threads and bone defect will be covered by autogenous bone graft and covered by titanium membrane.
  Osstell instrument will be used to measure and record fixture primary stability in ISQ units.
  Sutures will be placed. Sutures will be removed 7 days later. Immediate postoperative CBCT will be performed. Antibiotic (combination of 500mg amoxicillin and 125mg clavulanic acid) and analgesic and anti-inflammatory (Ibuprofen 600mg) will be prescribed.
  Interventions: Procedure: Autogenous bone for bone augmentation

INTERVENTIONS:
Procedure: Mineralized plasmatic matrix for bone augmentation — Vertical bone augmentation of defective posterior mandibular alveolar ridge using MPM (Mineralized Plasmatic Matrix) bone graft.
  Other Names: Sticky bone graft
  Arms: Interventional
Procedure: Autogenous bone for bone augmentation — Vertical bone augmentation of defective posterior mandibular alveolar ridge using autogenous bone graft (gold standard) covered by titanium membrane.
  Arms: Comparator

SUMMARY:
* Patients will be diagnosed to determine whether they are eligible for the inclusion criteria of this study or not. Patients who are eligible will start their surgical treatment in the next visit after radiographic and surgical site evaluation.
* On the day of surgery, each patient will be assigned to either intervention or control group, the patients will receive inferior alveolar nerve block and long buccal nerve anesthesia. Future implant site will be planned, an incision will be made and flap will be reflected along the defective ridge.
* Implant fixture/s will be inserted in the previously planned site. Uncovered fixture threads and bone defect will be covered by MPM or autogenous bone graft.
* In the control group, autogenous particulate bone graft will be used for vertical augmentation and covered with titanium reinforced membrane. In the intervention group, MPM (Mineralized plasmatic matrix) will be used.
* Edges will be approximated, Sutures will be placed.
* Osstell instrument will be used to measure and record fixture primary stability in ISQ units.
* Patients will be referred to the fixed prosthodontics department for placement of the crowns after ensuring success of osseointegration and implant stability (after 4 months).
* Patients will evaluate their overall satisfaction after fitting the final prosthesis using a questionnaire at 9 months.
* After 9 months, CBCT will be performed to evaluate augmented bone height to be compared with the bone height previously recorded in CBCT.
* Osstell instrument will be used to evaluate the implant stability ratio in ISQ unit to be compared to the ratio recorded before.

DETAILED DESCRIPTION:
In the study group:

* Full medical and dental history will be obtained from all the patients participating in this study (figure 2).
* Thorough clinical and radiographic examination for the ridge area to be treated will be done.
* Future implant site will be planned.
* Each patient will be asked to evaluate their overall satisfaction using a questionnaire before any intervention.
* Patients will receive 2 gm of amoxicillin 1 hour before surgery. They will be instructed to wash their mouths with a 0.12% chlorhexidine solution for 30 seconds immediately before surgery.
* The patient will receive inferior alveolar nerve block and long buccal nerve anesthesia using articane HCl 4% with 1:100,000 adrenaline local anesthetic solution using aspirating syringe and 27-gauge needle.
* After confirming the success of profound local anaesthesia, an incision will be made and flap will be reflected along the ridge of the previously planned intraoral donor site to completely expose bone.
* Autogenous bone graft will be obtained and will be grinded according to the dimensions of the present defect.
* MPM (Mineralized plasmatic matrix) will be prepared:

Tubes of 9 ml of venous blood will be taken from the patient and will be placed in a centrifuge at 2500 rpm / min for 5 min.

At the end of the centrifugation, the blood in the tube will be separated into two compartments one yellow and one red.

The yellow part will be withdrawn with a syringe to be mixed with the grinded autogenous bone previously obtained from intra oral site.

Components will be mixed using a probe until the formation of a single homogeneous component, called the MPM (Mineralized Plasmatic Matrix).

* The graft site receiver will be prepared by perforating the lateral cortical bone to improve the vascularization and facilitate cell migration.
* Implant fixture/s will be inserted in the previously planned site.
* Uncovered fixture threads and bone defect will be covered by MPM.
* Osstell instrument will be used to measure and record fixture primary stability in ISQ units precisely and objectively 48.
* Edges will be approximated, Sutures will be placed.
* Sutures will be removed 7 days later.
* Immediate postoperative CBCT will be performed.
* Antibiotic (combination of 500mg amoxicillin and 125mg clavulanic acid) and analgesic and anti-inflammatory (Ibuprofen 600mg) will be prescribed after the surgical procedure to be administrated by the patients.
* Patients will be referred to the fixed prosthodontics department for placement of the crowns after ensuring success of osseointegration and implant stability (after 4 months).

In the control group:

* The Same previously mentioned procedure will be performed, But here gold standards are to be performed (Autogenous particulate bone graft used for vertical augmentation will be covered with titanium reinforced membrane).
* Osstell tool will be used to measure and record fixture primary stability in ISQ units.
* Suturing will be performed.
* Then Immediate Post operative CBCT will be performed.
* Antibiotic (combination of 500mg amoxicillin and 125mg clavulanic acid) and analgesic and anti-inflammatory (Ibuprofen 600mg) will be prescribed after the surgical procedure to be administrated by the patients.
* Patients will be referred to the fixed prosthodontics department for placement of the crowns after ensuring success of osseointegration and implant stability (after 4 months).

Postoperative follow up in both groups:

* After 4 months, Osstell instrument will be used to evaluate the implant stability ratio in ISQ unit to be compared to the ratio recorded before.
* After 9 months, Patients will evaluate their overall satisfaction after fitting the final prosthesis using a questionnaire to be answered by YES or NO.
* -After 9 months, CBCT will be performed to evaluate augmented bone height to be compared with the bone height previously recorded in CBCT.

ELIGIBILITY:
Inclusion Criteria:

1. Medically free patients.
2. Patients with posterior mandibular defective partially edentulous ridge.
3. Evaluated bone height on CBCT to be (0-4 mm buccal bone dehiscence) and width (not less than 4.5 mm)
4. Patients physically able to tolerate surgical and restorative procedures.
5. Patients with an opposing tooth to the pre-implant site.
6. Good oral hygiene.
7. Highly motivated patients.

Exclusion Criteria:

1. Patients allergic to local anaesthetic agent.
2. smokers.
3. Pregnant or lactating females.
4. Presence of any pathosis in the pre-implant site.
5. Presence of parafunctional habits.
6. History of oral radiotherapy.
7. History of prolonged steroids use.
8. Psychological disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Implant body stability in ISQ unit | Change from baseline implant body stability at 4 months

SECONDARY OUTCOMES:
Bone height in Cone beam CT | Change from baseline bone height at 9 months

OTHER OUTCOMES:
Patient satisfaction using questionnare | 9 months

IPD SHARING:
Plan to Share IPD: No